CLINICAL TRIAL: NCT03802422
Title: Perineural Injection Therapy With Vitamin B12 for Carpal Tunnel Syndrome
Brief Title: Vitamin B12 for Carpal Tunnel Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It is hard to enroll patients due to Covid-19 pandemic.
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vitamin for CTS
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hydrodissection; Vitamin B12
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Vitamin B 12; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B12 hydrodissection (Experimental): Ultrasound-guided hydrodissection with Vitamin B12 between carpal tunnel and median nerve.
  Interventions: Drug: Vitamin B12
- Normal saline hydrodissection (Placebo Comparator): Ultrasound-guided hydrodissection with normal saline between carpal tunnel and median nerve.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Vitamin B12 — Ultrasound-guided hydrodissection with 3cc Vitamin B12 (methycobal, 500μg/ml) between carpal tunnel and median nerve.
  Arms: Vitamin B12 hydrodissection
Drug: Normal saline — Ultrasound-guided hydrodissection with 3cc 0.9% normal saline between carpal tunnel and median nerve.
  Arms: Normal saline hydrodissection

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. The hydrodissection could decrease the entrapment of nerve to restore blood supply. In addition, the Vitamin B12 was considered to be beneficial for peripheral neuropathy and pain relief. The investigators design a randomized, double-blind, controlled trail to assess the effect after ultrasound-guided hydrodissection with Vitamin B12 in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients with mild to moderate CTS will been randomized into intervention and control group. Participants in intervention group received one-dose ultrasound-guided hydrodissection with 3cc Vitamin B12 and control side received one-dose ultrasound-guided injection 3cc normal saline. No additional treatment after injection through the study period. The primary outcome is Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve. The evaluation was performed pretreatment as well as on the 2nd week, 1st, 2nd, 3rd and 6th month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd , 3rd and 6th month after injection
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd , 3rd and 6th month after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of electrophysiological measurement on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd , 3rd and 6th month after injection
  Antidromic sensory nerve conduction velocity of the median nerve before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Smith J, Wisniewski SJ, Finnoff JT, Payne JM. Sonographically guided carpal tunnel injections: the ulnar approach. J Ultrasound Med. 2008 Oct;27(10):1485-90. doi: 10.7863/jum.2008.27.10.1485. PMID 18809959
- [Result] Wu YT, Chen SR, Li TY, Ho TY, Shen YP, Tsai CK, Chen LC. Nerve hydrodissection for carpal tunnel syndrome: A prospective, randomized, double-blind, controlled trial. Muscle Nerve. 2019 Feb;59(2):174-180. doi: 10.1002/mus.26358. Epub 2018 Dec 4. PMID 30339737
- [Result] Wu YT, Ke MJ, Ho TY, Li TY, Shen YP, Chen LC. Randomized double-blinded clinical trial of 5% dextrose versus triamcinolone injection for carpal tunnel syndrome patients. Ann Neurol. 2018 Oct;84(4):601-610. doi: 10.1002/ana.25332. Epub 2018 Oct 4. PMID 30187524
- [Result] Xu G, Lv ZW, Feng Y, Tang WZ, Xu GX. A single-center randomized controlled trial of local methylcobalamin injection for subacute herpetic neuralgia. Pain Med. 2013 Jun;14(6):884-94. doi: 10.1111/pme.12081. Epub 2013 Apr 8. PMID 23566267